CLINICAL TRIAL: NCT04813484
Title: Addressing Violence and HIV Cascade of Care Outcomes Among Transgender Women
Brief Title: Addressing Violence and HIV Care Among Transgender Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Kristi Gamarel, Associate Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: F056257; R21MH121974 (NIH)
Record Dates: First submitted 2021-03-21; First posted 2021-03-24 (Actual); Results first posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Acceptability of Health Care; HIV Infections
MeSH Terms: conditions — Patient Acceptance of Health Care; HIV Infections

STUDY DESIGN:
Intervention Model Description: One-arm pilot
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Kicking it with the Gurlz (Experimental): This multicomponent intervention includes a violence and gender affirmation screening tool, a peer delivered adaptation of the group-level Seeking Safety Program, and individual-level peer navigation sessions.
  Interventions: Behavioral: Kickin it with the Gulz

INTERVENTIONS:
Behavioral: Kickin it with the Gulz — The intervention is a multicomponent intervention, including a screening, groups, and individual sessions.

SUMMARY:
This project seeks to adapt and pilot a trauma-informed combination intervention named 'Kickin' it with the Gurlz' that was designed with, for, and by transgender women of color to improve HIV care continuum outcomes. The intervention components include a violence and gender affirmation screening tool, a peer-led adaptation of Seeking Safety, and individual-level peer navigation sessions. The project will examine the feasibility, acceptability, and preliminary promise of the multicomponent by conducting a one-arm pilot with 30 transgender women of color who have a history of trauma. Participants will complete baseline, immediate post-intervention, and 3-month follow up assessments.

DETAILED DESCRIPTION:
This project seeks to evaluate the feasibility and acceptability of the trauma-informed combination care intervention to improve HIV care continuum outcomes including the development of community-informed strategies for subsequent RCTs. We will conduct a one-arm pilot of the adapted multicomponent trauma-informed intervention named "Kickin it with the Gurlz." This project will collect feasibility and acceptability data related to identifying, recruiting, enrolling, intervening with, and retaining participants (i.e. recruitment length, screening procedures, feasibility of conducting sessions, intervention acceptability, retention rates, feasibility of verifying self-reported and medical chart review data on viral load and exit interviews with participants and staff at program conclusion). The study will recruit 30 participants into the pilot study. Participants will complete baseline, end of program, and 3-month post-intervention follow-up surveys. Exit interviews and interviews with key stakeholders will identify strategies for implementing trauma-informed HIV treatment efficacy trials with transgender women of color within close-knit communities, such as acceptable and feasible control conditions, acceptable and feasible violence and gender affirmation screening, biomedical confirmation methods, contamination concerns, and potential changes needed within existing health care systems.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Assigned male at birth; identifies as female, transgender woman, or another feminine gender identity
* Self-identifies as a person of color (any racial/ethnic identity except non-Hispanic white)
* Self-reports as HIV-positive
* History of trauma (i.e., endorses at least 2 items on the adapted Trauma History Screener which includes IPV and experiencing or witnessing other forms of violence for transgender women
* Living or willing to travel to Detroit
* English-speaking
* Willing and able to provide informed consent.

Exclusion Criteria:

• Evidence of severe cognitive impairment or active psychosis that may impede ability to provide fully informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — All participants will identify their gender as a female, transgender woman, or another feminine gender identity.
Enrollment: 11 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristi Gamarel, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
Our team is committed to collaboration with NIH officials, other researchers, the health and social services community, and other entities for rapid dissemination of data and sharing of materials. We will make our results available to the community of researchers and general public interested in transgender health to avoid unintentional duplication of research, as well as to others in the health and social services community, including HIV clinics, LGBT community based organizations, and AIDS service organizations.

RESULTS

PARTICIPANT FLOW:
Groups:
- Kicking it With the Gurlz: This multicomponent intervention includes a violence and gender affirmation screening tool, a peer delivered adaptation of the group-level Seeking Safety Program, and individual-level peer navigation sessions.
  Kickin it with the Gurlz: This multicomponent intervention includes a violence and gender affirmation screening tool, a peer delivered adaptation of the group-level Seeking Safety Program, and individual-level peer navigation sessions.
Period: Overall Study
Arm/Group | Kicking it With the Gurlz
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Kicking it With the Gurlz
Number analyzed (Participants) | 11
Age, Continuous [Mean (Full Range); unit: years] | 29 [19 to 41]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Acceptability Quantitative
Description: The Client Satisfaction Questionnaire (CSQ-8) will be used to assess intervention satisfaction. Scores are averaged across items once. Items 2, 4, 5, and 8 are reverse scored. Total scores range from 0 to 4, with the higher number indicating greater satisfaction.
Time Frame: 3-month follow up
Population: Descriptive analyses examining the mean.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Kicking it With the Gurlz
Number analyzed (Participants) | 11
score on a scale | 3.5 [0 to 4]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Kicking it With the Gurlz
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/84/NCT04813484/Prot_001.pdf
  • Informed Consent Form (2021-06-28): https://cdn.clinicaltrials.gov/large-docs/84/NCT04813484/ICF_002.pdf